CLINICAL TRIAL: NCT04628585
Title: Long-term Follow-up of Subjects with Sickle Cell Disease Treated with Ex Vivo Gene Therapy Using Autologous Hematopoietic Stem Cells Transduced with a Lentiviral Vector
Brief Title: Long-term Follow-up of Subjects with Sickle Cell Disease Treated with Ex Vivo Gene Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-307; 2019-004266-18 (EudraCT Number); 2024-513901-30-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Sickle Cell Disease
Keywords: Hematopoietic Stem Cells
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Safety

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subjects with sickle-cell disease: Subjects treated with ex vivo gene therapy drug product for sickle cell disease in a bluebird bio-sponsored study who agree to participate in this long-term follow-up study
  Interventions: Other: Safety and efficacy assessments

INTERVENTIONS:
Other: Safety and efficacy assessments — Safety evaluations, disease-specific assessments, and assessments to monitor for long-term complications of autologous transplant

SUMMARY:
This is a multi-center, long-term safety and efficacy follow-up study for subjects with sickle cell disease who have been treated with ex vivo gene therapy drug product in bluebird bio-sponsored clinical studies. After completing the parent clinical study (approximately 2 years), eligible subjects will be followed for an additional 13 years for a total of 15 years post-drug product infusion. No investigational drug product will be administered in the study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for this study by subject, or as applicable, subject's parent(s)/legal guardian(s)
* Treated with drug product for therapy of sickle cell disease in a bluebird bio-sponsored clinical study

Exclusion Criteria:

* There are no exclusion criteria for this study

Ages: 2 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with sickle cell disease treated with ex vivo gene therapy product in bluebird bio-sponsored clinical studies
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2038-01 (Estimated); Study Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with immune-related AEs (e.g., autoimmune disorders, GVHD, opportunistic infections, HIV) | Through 15 years post-drug product infusion
Number of subjects with new or worsening hematologic disorders | Through 15 years post-drug product infusion
Number of subjects with new or worsening neurologic disorders | Through 15 years post-drug product infusion
Number of subjects with malignancies | Through 15 years post-drug product infusion

SECONDARY OUTCOMES:
Proportion of subjects with complete resolution of severe VOEs (sVOE-CR) over time through Year 15 | Through 15 years post-drug product infusion
Proportion of subjects with complete resolution of VOEs (VOE-CR) over time through Year 15 | Through 15 years post-drug product infusion
Annualized number of severe VOEs over time through Year 15 | Through 15 years post-drug product infusion
Annualized number of VOEs over time through Year 15 | Through 15 years post-drug product infusion
Change from parent study baseline in annualized number of severe VOEs over time through Year 15 | Through 15 years post-drug product infusion
Assessment of total Hb over time post-drug product infusion through Year 15 | Through 15 years post-drug product infusion
Assessment of non-transfused total Hb over time post-drug product infusion through Year 15 | Through 15 years post-drug product infusion
  Non-transfused total Hb refers to the total g/dL of HbS + HbF + HbA2 + HbAT87Q
Assessment of HbS percentage of non-transfused total Hb over time post-drug product infusion through Year 15 | Through 15 years post-drug product infusion
  Non-transfused total Hb refers to the total g/dL of HbS + HbF + HbA2 + HbAT87Q
Assessment of HbAT87Q percentage of non-transfused total Hb over time post-drug product infusion through Year 15 | Through 15 years post-drug product infusion
  Non-transfused total Hb refers to the total g/dL of HbS + HbF + HbA2 + HbAT87Q
Assessment of non-HbS percentage of non-transfused total Hb over time post-drug product infusion through Year 15 | Through 15 years post-drug product infusion
  Non-transfused total Hb refers to the total g/dL of HbS + HbF + HbA2 + HbAT87Q. Non-HbS is the total g/dL of HbF + HbA2 + HbAT87Q
Change from parent study baseline through Year 15 in hemolysis markers | Through 15 years post-drug product infusion
  Change from parent study baseline through Year 15 in absolute reticulocyte count, percent reticulocytes/erythrocytes, total bilirubin, indirect bilirubin, haptoglobin, and lactate dehydrogenase hemolysis markers
Change from parent study baseline through Year 15 in markers of iron stores | 15 years post-drug product infusion
  Change from parent study baseline through Year 15 in serum ferritin and liver iron content markers of iron stores

CONTACTS AND LOCATIONS:
Overall Officials: Anjulika Chawla, MD, Study Director — bluebird bio, Inc.
Locations (16):
- United States (15):
  - University of Alabama, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Hospital Necker, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Bluebird bio is committed to transparency. Appropriately de-identified patient-level datasets and supporting documents may be shared (if contractually or otherwise legally permitted) following study completion and once all applicable regulatory submissions based on this study have been performed. Sharing of individual patient data will be done according to criteria established by bluebird bio and/or industry best practices to protect confidential information and maintain the privacy of study participants. For inquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Magrin E, Semeraro M, Hebert N, Joseph L, Magnani A, Chalumeau A, Gabrion A, Roudaut C, Marouene J, Lefrere F, Diana JS, Denis A, Neven B, Funck-Brentano I, Negre O, Renolleau S, Brousse V, Kiger L, Touzot F, Poirot C, Bourget P, El Nemer W, Blanche S, Treluyer JM, Asmal M, Walls C, Beuzard Y, Schmidt M, Hacein-Bey-Abina S, Asnafi V, Guichard I, Poiree M, Monpoux F, Touraine P, Brouzes C, de Montalembert M, Payen E, Six E, Ribeil JA, Miccio A, Bartolucci P, Leboulch P, Cavazzana M. Long-term outcomes of lentiviral gene therapy for the beta-hemoglobinopathies: the HGB-205 trial. Nat Med. 2022 Jan;28(1):81-88. doi: 10.1038/s41591-021-01650-w. Epub 2022 Jan 24. PMID 35075288
- See also: HGB-205 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT02151526?term=HGB-205&cond=Sickle+Cell+Disease&draw=2&rank=1
- See also: HGB-206 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT02140554?term=HGb-206&cond=Sickle+Cell+Disease&draw=2&rank=1
- See also: HGB-210 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT04293185?term=HGB-210&cond=Sickle+Cell+Disease&draw=2&rank=1